CLINICAL TRIAL: NCT02019420
Title: A Phase 3 Randomized Double-blind Study Comparing TR-701 FA and Linezolid in Ventilated Gram-positive Nosocomial Pneumonia
Brief Title: Tedizolid Phosphate (TR-701 FA, MK-1986) vs Linezolid for the Treatment of Nosocomial Pneumonia (MK-1986-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1986-002; TR701-132 (Other: Cubist Protocol Number); 2013-004154-22 (EudraCT Number); MK-1986-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — tedizolid phosphate; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Tedizolid phosphate IV (Experimental): Ventilated HABP/VABP participants receive tedizolid phosphate 200 mg IV once daily for 7 days, or for 14 days for concurrent bacteremia.
  Interventions: Drug: Tedizolid phosphate
- Linezolid IV (Active Comparator): Ventilated HABP/VABP participants receive linezolid 600 mg IV every 12 hours for 10 days, or for 14 days for concurrent bacteremia.
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Tedizolid phosphate — Tedizolid phosphate IV 200 mg once daily
  Other Names: SIVEXTRO®; TR-701 FA; MK-1986
  Arms: Tedizolid phosphate IV
Drug: Linezolid — Linezolid IV 600 mg twice daily
  Other Names: ZYVOX®
  Arms: Linezolid IV

SUMMARY:
This is a 1:1 ratio, randomized, double-blind, double-dummy, multicenter, global Phase 3 study of tedizolid phosphate (TR-701 FA) 200 mg intravenous (IV) once daily for 7 days versus linezolid (Zyvox®, Zyvoxid®, etc) 600 mg IV every 12 hours for 10 days for the treatment of ventilated participants with presumed gram-positive hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP), collectively referred to as ventilated nosocomial pneumonia (VNP). Participants with concurrent gram-positive bacteremia are to receive 14 days of active therapy in either treatment arm.

The primary objective is to determine the noninferiority (NI) in all-cause mortality (ACM) within 28 days after randomization of IV tedizolid phosphate compared with IV linezolid in the Intent to Treat (ITT) Analysis Set (NI is declared when the lower bound of the 95% CI > -10).

ELIGIBILITY:
Inclusion Criteria:

* Requires IV antibiotic therapy with diagnosis of ventilated nosocomial pneumonia
* Gram-positive bacteria on respiratory Gram stain

Exclusion Criteria:

* Pneumonia of community, viral, fungal or parasitic etiology
* Structural lung abnormalities
* Immunosuppression
* Previous antibiotics for > 24 hours
* Expected survival of < 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Alp E, Voss A. Ventilator associated pneumonia and infection control. Ann Clin Microbiol Antimicrob. 2006 Apr 6;5:7. doi: 10.1186/1476-0711-5-7. PMID 16600048
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] Lan KK, Wittes J. The B-value: a tool for monitoring data. Biometrics. 1988 Jun;44(2):579-85. PMID 3390511
- [Background] Lawrence KR, Adra M, Gillman PK. Serotonin toxicity associated with the use of linezolid: a review of postmarketing data. Clin Infect Dis. 2006 Jun 1;42(11):1578-83. doi: 10.1086/503839. Epub 2006 Apr 27. PMID 16652315
- [Background] Lemaire S, Van Bambeke F, Appelbaum PC, Tulkens PM. Cellular pharmacokinetics and intracellular activity of torezolid (TR-700): studies with human macrophage (THP-1) and endothelial (HUVEC) cell lines. J Antimicrob Chemother. 2009 Nov;64(5):1035-43. doi: 10.1093/jac/dkp267. Epub 2009 Sep 16. PMID 19759040
- [Background] Torres A, Ewig S, Lode H, Carlet J; European HAP working group. Defining, treating and preventing hospital acquired pneumonia: European perspective. Intensive Care Med. 2009 Jan;35(1):9-29. doi: 10.1007/s00134-008-1336-9. Epub 2008 Nov 7. PMID 18989656
- [Background] Drusano GL, Liu W, Kulawy R, Louie A. Impact of granulocytes on the antimicrobial effect of tedizolid in a mouse thigh infection model. Antimicrob Agents Chemother. 2011 Nov;55(11):5300-5. doi: 10.1128/AAC.00502-11. Epub 2011 Sep 12. PMID 21911576
- [Background] Garonzik SM, Li J, Thamlikitkul V, Paterson DL, Shoham S, Jacob J, Silveira FP, Forrest A, Nation RL. Population pharmacokinetics of colistin methanesulfonate and formed colistin in critically ill patients from a multicenter study provide dosing suggestions for various categories of patients. Antimicrob Agents Chemother. 2011 Jul;55(7):3284-94. doi: 10.1128/AAC.01733-10. Epub 2011 May 9. PMID 21555763
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children: executive summary. Clin Infect Dis. 2011 Feb 1;52(3):285-92. doi: 10.1093/cid/cir034. PMID 21217178
- [Background] Pletz MW, Burkhardt O, Welte T. Nosocomial methicillin-resistant Staphylococcus aureus (MRSA) pneumonia: linezolid or vancomycin? - Comparison of pharmacology and clinical efficacy. Eur J Med Res. 2010 Nov 30;15(12):507-13. doi: 10.1186/2047-783x-15-12-507. PMID 21163725
- [Background] Tessier PR, Keel RA, Hagihara M, Crandon JL, Nicolau DP. Comparative in vivo efficacies of epithelial lining fluid exposures of tedizolid, linezolid, and vancomycin for methicillin-resistant Staphylococcus aureus in a mouse pneumonia model. Antimicrob Agents Chemother. 2012 May;56(5):2342-6. doi: 10.1128/AAC.06427-11. Epub 2012 Feb 21. PMID 22354302
- [Background] Wunderink RG, Niederman MS, Kollef MH, Shorr AF, Kunkel MJ, Baruch A, McGee WT, Reisman A, Chastre J. Linezolid in methicillin-resistant Staphylococcus aureus nosocomial pneumonia: a randomized, controlled study. Clin Infect Dis. 2012 Mar 1;54(5):621-9. doi: 10.1093/cid/cir895. Epub 2012 Jan 12. PMID 22247123
- [Derived] Mikamo H, Nagashima M, Kusachi S, Fujimi S, Oshima N, De Anda C, Takase A. Efficacy and safety of tedizolid for the treatment of ventilated gram-positive hospital-acquired or ventilator-associated bacterial pneumonia in Japanese patients: Results from a subgroup analysis of a phase 3, randomized, double-blind study comparing tedizolid and linezolid. J Infect Chemother. 2022 Sep;28(9):1235-1241. doi: 10.1016/j.jiac.2022.04.027. Epub 2022 Jun 16. PMID 35718656
- [Derived] Wunderink RG, Roquilly A, Croce M, Rodriguez Gonzalez D, Fujimi S, Butterton JR, Broyde N, Popejoy MW, Kim JY, De Anda C. A Phase 3, Randomized, Double-Blind Study Comparing Tedizolid Phosphate and Linezolid for Treatment of Ventilated Gram-Positive Hospital-Acquired or Ventilator-Associated Bacterial Pneumonia. Clin Infect Dis. 2021 Aug 2;73(3):e710-e718. doi: 10.1093/cid/ciab032. PMID 33720350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ventilated participants with presumed gram-positive hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP) were enrolled at study sites located in 34 countries.
Groups:
- Tedizolid: Ventilated HABP/VABP participants received tedizolid phosphate 200 mg IV once daily for 7 days, or for 14 days for concurrent bacteremia.
- Linezolid: Ventilated HABP/VABP participants received linezolid 600 mg IV every 12 hours for 10 days, or for 14 days for concurrent bacteremia.
Period: Overall Study
Arm/Group | Tedizolid | Linezolid
Started (Randomized) | 366 | 360
Treated | 361 | 357
Completed | 258 | 254
Not Completed | 108 | 106
Not completed — Did not receive study drug | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — At request of sponsor or investigator | 0 | 1
Not completed — Death | 104 | 99
Not completed — Transferred to other care facility | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tedizolid | Linezolid | Total
Number analyzed (Participants) | 366 | 360 | 726
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (18.41) | 58.7 (17.44) | 58.4 (17.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 106 | 223
  Male | 249 | 254 | 503
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 61 | 126
  Not Hispanic or Latino | 290 | 289 | 579
  Unknown or Not Reported | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 68 | 70 | 138
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 11 | 14
  White | 269 | 258 | 527
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality in the Intent-to-Treat (ITT) Population
Description: The numbers of participants with all-cause mortality within 28 days after randomization was determined in the ITT population. Any participants who were lost to follow-up and not known to be alive or deceased by Day 28 were imputed as deceased.
Time Frame: Up to 28 days
Population: The ITT set is all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 366 | 360
Participants | 103 | 95
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Non-Inferiority — Difference in ITT all-cause mortality (linezolid - tedizolid). Noninferiority is declared when the lower bound of the 95% CI > -10; Difference in all-cause mortality = -1.8, 95% CI 2-sided [-8.2 to 4.7] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

2. Secondary Outcome: Number of Participants With All-Cause Mortality in the Microbiological Intent-to-Treat (mITT) Population
Description: The numbers of participants with all-cause mortality within 28 days after randomization was determined in the mITT population. Any participants who were lost to follow-up and not known to be alive or deceased by Day 28 were imputed as deceased.
Time Frame: Up to 28 days
Population: The mITT set is all randomized, treated participants who have gram-positive pathogen(s) confirmed by respiratory tract/pleural fluid culture results obtained within 36 hours (or 72 hours if methicillin-resistant S. aureus [MRSA]) before first study drug dose, and bacterial pathogen against which the investigational drug has antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 178 | 202
Participants | 46 | 49
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in mITT all-cause mortality (linezolid - tedizolid); Difference in all-cause mortality = -1.6, 95% CI 2-sided [-10.3 to 7.1] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

3. Secondary Outcome: Clinical Response at Test of Cure (TOC) Visit in the Intent-to-Treat (ITT) Population
Description: The clinical response in the ITT population at the TOC visit (derived from the Investigator's assessment at the EOT and TOC visits) was determined by the investigator to be either: clinical success, clinical failure, or indeterminate. Clinical success was declared when most or all clinical signs were completely resolved, with no new signs of infection, no additional antibiotic therapy was required, and the participant was alive. Indeterminate was declared when the investigator could not determine success or failure. Clinical failure was declared with progression, relapse, or recurrence of new symptoms of infection, or a persistence or insufficient improvement in signs and symptoms of VNP.
Time Frame: 7-14 days after end of therapy - TOC
Population: The ITT set includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 366 | 360
Participants
  Clinical Success | 206 | 230
  Clinical Failure | 144 | 110
  Indeterminate | 16 | 20
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in ITT clinical success (tedizolid - linezolid); Difference in clinical success = -7.6, 95% CI 2-sided [-14.7 to -0.5] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

4. Secondary Outcome: Clinical Response at Test of Cure (TOC) Visit in the Clinically-Evaluable (CE) Population
Description: The clinical response in the CE population at the TOC visit (derived from the Investigator's assessment at the EOT and TOC visits) was determined by the investigator to be either: clinical success, clinical failure, or indeterminate. Clinical success was declared when most or all clinical signs were completely resolved, with no new signs of infection, no additional antibiotic therapy was required, and the participant was alive. Indeterminate was declared when the investigator could not determine success or failure. Clinical failure was declared with progression, relapse, or recurrence of new symptoms of infection, or a persistence or insufficient improvement in signs and symptoms of VNP.
Time Frame: 7-14 days after end of therapy - TOC
Population: The CE set is all randomized and treated participants who had assessment data available and did not have confounding events.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 267 | 243
Participants
  Clinical Success | 143 | 146
  Clinical Failure | 124 | 97
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in CE clinical success (tedizolid - linezolid); Difference in clinical success = -6.5, 95% CI 2-sided [-15.1 to 2.1] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

5. Secondary Outcome: Number of Methicillin-Susceptible Staphylococcus Aureus (MSSA)-Infected Participants With All-Cause Mortality in the Microbiological Intent-to-Treat (mITT) Population
Description: The number of MSSA-infected participants with all-cause mortality within 28 days after randomization was determined in the mITT population. Participants who had confirmed MSSA culture results from respiratory tract or pleural fluid specimens obtained within 36 hours of study Day 1 were included. Any participants who were lost to follow-up and not known to be alive or deceased by Day 28 were imputed as deceased.
Time Frame: Up to 28 days
Population: The MSSA-infected mITT set is all randomized, treated participants who have MSSA confirmed by respiratory tract/pleural fluid culture results obtained within 36 hours before first study drug dose, and documented bacterial pathogen against which the investigational drug has antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 117 | 128
Participants | 31 | 32
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in MSSA mITT all-cause mortality (linezolid - tedizolid); Difference in all-cause mortality = -1.5, 95% CI 2-sided [-12.5 to 9.5] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

6. Secondary Outcome: Number of Methicillin-Resistant Staphylococcus Aureus (MRSA)-Infected Participants With All-Cause Mortality in the Microbiological Intent-to-Treat (mITT) Population
Description: The number of MRSA-infected participants with all-cause mortality within 28 days after randomization was determined in the mITT population. Participants who had confirmed MRSA culture results from respiratory tract or pleural fluid specimens obtained within 72 hours of study Day 1 were included. Any participants who were lost to follow-up and not known to be alive or deceased by Day 28 were imputed as deceased.
Time Frame: Up to 28 days
Population: The MRSA-infected mITT set is all randomized, treated participants who have MRSA confirmed by respiratory tract/pleural fluid culture results obtained within 72 hours before first study drug dose, and documented bacterial pathogen against which the investigational drug has antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 54 | 69
Participants | 14 | 20
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in MRSA mITT all-cause mortality (linezolid - tedizolid); Difference in all-cause mortality = 3.1, 95% CI 2-sided [-12.8 to 18.9] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

7. Secondary Outcome: Number of Participants With a Favorable Response at End-of-Therapy (EOT) Visit in the Microbiological Intent-to-Treat (mITT) Population
Description: The number of patients in the mITT population with a favorable response at EOT was determined. Favorable response included eradication (absence of the baseline pathogen) and presumed eradication (no source specimen to culture in a participant assessed as a clinical cure by the investigator).
Time Frame: 1-3 days after completing study therapy (Days 8-10 or Days 15-17)
Population: The mITT set is all randomized, treated participants who have gram-positive pathogen(s) confirmed by respiratory tract/pleural fluid culture results obtained within 36 hours (or 72 hours if MRSA) before first study drug dose, and documented bacterial pathogen against which the investigational drug has antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 178 | 202
Participants | 123 | 166
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in mITT favorable response (tedizolid - linezolid); Difference in clinical success = -13.1, 95% CI 2-sided [-21.7 to -4.5] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

8. Secondary Outcome: Number of Participants With a Favorable Response at End-of-Therapy (EOT) Visit in the Microbiologically-Evaluable 1 (ME-1) Population
Description: The number of patients in the ME-1 population with a favorable response at EOT was determined. Favorable response included eradication (absence of the baseline pathogen) and presumed eradication (no source specimen to culture in a participant assessed as a clinical cure by the investigator).
Time Frame: 1-3 days after completing study therapy (Days 8-10 or Days 15-17)
Population: The ME-1 set is all mITT participants who did not receive an antibiotic (other than study drug) with activity against the baseline pathogen up to 28 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 178 | 202
Participants | 123 | 166
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in ME-1 favorable response (tedizolid - linezolid); Difference in clinical success = -13.1, 95% CI 2-sided [-21.7 to -4.5] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

9. Secondary Outcome: Number of Participants With a Favorable Response at Test-of-Cure (TOC) Visit in the Microbiological Intent-to-Treat (mITT) Population
Description: The number of patients in the mITT population with a favorable response at TOC was determined. Favorable response included eradication (absence of the baseline pathogen) and presumed eradication (no source specimen to culture in a participant assessed as a clinical cure by the investigator).
Time Frame: 7-14 days after end of therapy - TOC
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 178 | 202
Participants | 117 | 158
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in mITT favorable response (tedizolid - linezolid); Difference in clinical success = -12.5, 95% CI 2-sided [-21.5 to -3.5] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

10. Secondary Outcome: Number of Participants With a Favorable Response at Test-of-Cure (TOC) Visit in the Microbiologically-Evaluable 2 (ME-2) Population
Description: The number of patients in the ME-2 population with a favorable response at TOC was determined. Favorable response included eradication (absence of the baseline pathogen) and presumed eradication (no source specimen to culture in a participant assessed as a clinical cure by the investigator).
Time Frame: 7-14 days after end of therapy - TOC
Population: The ME-2 set is all mITT participants who did not receive an antibiotic (other than study drug) with activity against the baseline pathogen up to the TOC visit and is also in the clinically-evaluable (CE) set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 120 | 109
Participants | 65 | 74
Statistical Analysis 1: Comparison: Tedizolid vs Linezolid; Test type: Other — Difference in ME-2 favorable response (tedizolid - linezolid); Difference in clinical success = -13.7, 95% CI 2-sided [-26.2 to -1.2] — Difference and 95% CI were calculated with the Miettinen and Nurminen method without stratification

11. Secondary Outcome: Number of Participants With ≥1 Adverse Events (AEs)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Safety analysis is based on actual treatment received instead of randomization.
Time Frame: Up to 32 days
Population: The safety set is all randomized participants who received any amount of study drug. A total of 4 participants were randomized to tedizolid but received linezolid.
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 357 | 361
Participants | 327 | 325

12. Secondary Outcome: Number of Participants Discontinuing Study Therapy Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Safety analysis was based on actual treatment received and not randomization.
Time Frame: Up to 14 days
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tedizolid | Linezolid
Number analyzed (Participants) | 357 | 361
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Up to 32 days
Description: All participants who received any amount of study drug are included. The safety assessment is based on actual treatment received, and thus the linezolid arm includes 4 participants randomized to tedizolid who received the wrong treatment.
Arm/Group | Tedizolid | Linezolid
All-Cause Mortality (participants affected / at risk) | 101/357 | 103/361
Serious Adverse Events (participants affected / at risk) | 129/357 | 149/361
Other Adverse Events (participants affected / at risk) | 176/357 | 175/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tedizolid (N=357) | Linezolid (N=361)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 21 (24) | 16 (16)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 7 (8) | 6 (6)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) | 3 (3)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossoptosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 8 (8) | 12 (12)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
CNS ventriculitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endotoxaemia (Infections and infestations) | 0 (0) | 1 (1)
Endotoxic shock (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 4 (4)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 6 (6)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Postoperative wound infection (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 6 (6) | 5 (5)
Septic shock (Infections and infestations) | 16 (16) | 18 (18)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Toxic shock syndrome (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Propofol infusion syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Benign enlargement of the subarachnoid spaces (Nervous system disorders) | 0 (0) | 1 (1)
Brain hypoxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 13 (13) | 7 (7)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral vasoconstriction (Nervous system disorders) | 0 (0) | 1 (1)
Cholinergic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis crisis (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 2 (2) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 7 (7)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tedizolid (N=357) | Linezolid (N=361)
Anaemia (Blood and lymphatic system disorders) | 56 (66) | 51 (52)
Constipation (Gastrointestinal disorders) | 31 (33) | 28 (31)
Diarrhoea (Gastrointestinal disorders) | 34 (36) | 49 (52)
Vomiting (Gastrointestinal disorders) | 19 (19) | 15 (16)
Urinary tract infection (Infections and infestations) | 26 (26) | 20 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 38 (49) | 34 (38)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 22 (26) | 26 (31)
Hypertension (Vascular disorders) | 19 (20) | 14 (14)
Hypotension (Vascular disorders) | 27 (28) | 25 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Cubist intends to pursue publication of the results of the study in cooperation with a lead Investigator, subject to the terms and conditions of the clinical study agreement between Cubist and Investigators. Cubist approval in writing is required for publication of any data subsets.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02019420/Prot_SAP_000.pdf